CLINICAL TRIAL: NCT00929591
Title: Phase III Comparison of Adjuvant Chemoendocrine Therapy With CAF and Concurrent or Delayed Tamoxifen to Tamoxifen Alone in Postmenopausal Patients With Involved Axillary Lymph Nodes and Positive Receptors
Brief Title: SWOG-8814 Tamoxifen With or Without Combination Chemotherapy in Postmenopausal Women Who Have Undergone Surgery for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000075692; U10CA032102 (NIH); SWOG-8814 (Other: SWOG); CAN-NCIC-MA9 (Other: NCIC-CTG); CLB-9194 (Other: CALGB); EST-4188 (Other: ECOG); NCCTG-883051 (Other: NCCTG); INT-0100 (Other: CTEP)
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Fluorouracil; Tamoxifen; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tamoxifen for five years (Active Comparator): tamoxifen for five years
  Interventions: Drug: endocrine therapy; Drug: tamoxifen citrate; Radiation: brachytherapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy
- CAF followed by tamoxifen for five years (Experimental): intermittent CAF X 6 courses followed by tamoxifen for five years
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: endocrine therapy; Drug: endocrine-modulating drug therapy; Drug: fluorouracil; Drug: tamoxifen citrate; Radiation: brachytherapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy
- CAF with concurrent tamoxifen for five years (Experimental): intermittent CAF X 6 courses with concurrent tamoxifen for five years
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: endocrine therapy; Drug: endocrine-modulating drug therapy; Drug: fluorouracil; Drug: tamoxifen citrate; Radiation: brachytherapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
  Arms: CAF followed by tamoxifen for five years; CAF with concurrent tamoxifen for five years
Drug: doxorubicin hydrochloride
  Arms: CAF followed by tamoxifen for five years; CAF with concurrent tamoxifen for five years
Drug: endocrine therapy
Drug: endocrine-modulating drug therapy
  Arms: CAF followed by tamoxifen for five years; CAF with concurrent tamoxifen for five years
Drug: fluorouracil
  Arms: CAF followed by tamoxifen for five years; CAF with concurrent tamoxifen for five years
Drug: tamoxifen citrate
Radiation: brachytherapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving tamoxifen alone is more effective in treating breast cancer than giving tamoxifen together with chemotherapy or after chemotherapy.

PURPOSE: This randomized phase III trial is studying giving tamoxifen with or without combination chemotherapy to compare how well they work in treating postmenopausal women who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare disease-free survival and overall survival of postmenopausal women with node-positive, estrogen and/or progesterone receptor-positive adenocarcinoma of the breast randomly assigned to postoperative adjuvant treatment with long-term (5 years) tamoxifen vs. CAF (cyclophosphamide/doxorubicin/fluorouracil) plus concurrent and long-term tamoxifen vs. CAF followed by long-term tamoxifen. II. Compare the relative toxicities of these three regimens.

OUTLINE: Randomized study. All patients are randomized on Arms I, II, and III. Lumpectomy patients must receive radiotherapy on Regimen A. At the discretion of the physician, mastectomy patients may receive radiotherapy on Regimen B for a tumor greater than 5 cm in diameter, 4 or more positive nodes, or extranodal extension of the tumor into the axillary fat. Patients randomized to Arm I who are to receive radiotherapy should begin as soon as feasible postoperatively; these patients may be irradiated while receiving tamoxifen. Patients on Arms II and III who are to receive radiotherapy are treated either postoperatively prior to registration or after completion of and recovery from 6 courses of CAF. Arm I: Antiestrogen Therapy. Tamoxifen, TMX, NSC-180973. Arm II: 3-Drug Combination Chemotherapy followed by Antiestrogen Therapy. CAF: Cyclophosphamide, CTX, NSC-26271; Doxorubicin, DOX, NSC-123127; Fluorouracil, 5-FU, NSC-19893; followed by TMX. Arm III: 3-Drug Combination Chemotherapy plus Concurrent Antiestrogen Therapy. CAF; plus concurrent TMX. Regimen A: Radiotherapy. Irradiation of the breast and underlying chest wall and (optionally) of the supraclavicular area and, if indicated, the axilla, using megavoltage equipment with photon energies of up to 6 MV followed, if indicated, by a tumor bed boost using either electrons or iridium-192 (192-Ir) implants. Regimen B: Radiotherapy. Irradiation of the chest wall using either megavoltage photons via a tangential field or electrons via a direct field plus (optional) photon irradiation of the supraclavicular area and, if indicated, the axilla.

PROJECTED ACCRUAL: 350 patients will be randomized to Arm I and 530 patients each will be randomized to Arms II and III. Accrual should be completed in about 4 years, and 4 additional years will be required for follow-up.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the breast No apocrine, adenoidcystic, or squamous carcinomas or sarcomas Pathologic Stage T1-3a, pathologic N1-2 (clinical N0-1), M0: Rendered free of gross tumor at surgery Primary tumor movable with respect to chest wall Axillary nodes movable with respect to chest wall and each other No preoperative edema of the arm, peau d'orange, skin ulceration, or inflammatory lesions One or more positive lymph nodes required No positive deep mastectomy margins or clinical skin involvement (focal microscopic dermal invasion or focal microscopic dermal lymphatic involvement allowed) No evidence of metastatic disease on pretherapy studies (including chest x-ray, bone scan, and mammogram) No bilateral invasive tumors Patients who had noninvasive ductal carcinoma in situ of the opposite breast and underwent prophylactic contralateral mastectomy are eligible Hormone receptor status: Positive for estrogen and/or progesterone receptors (at least 10 fmol/mg protein or unequivocally positive immunocytochemical assay for one or both) Participation in SWOG-8854 (flow cytometry) recommended

PATIENT CHARACTERISTICS: Age: Any age Sex: Females only Menopausal status: Postmenopausal as defined by 1 or more of the following: Bilateral oophorectomy at least 2 months prior to diagnosis of breast cancer (with or without estrogen therapy following surgery) Prior hysterectomy with at least 1 ovary remaining and either over 60 years old or with a postmenopausal FSH level Natural menopause (last menstrual period at least 1 year prior to registration or 4-12 months prior to registration with a postmenopausal FSH level) Treated with postmenopausal estrogen therapy and either over 55 years old or with a postmenopausal FSH level Performance status: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no more than 1.2 x normal Alkaline phosphatase no more than 1.2 x normal SGOT or SGPT no more than 1.2 x normal Renal: Creatinine no more than 2.0 mg/dL Cardiovascular: No uncontrolled hypertension No history of ischemic heart disease or CHF Normal ejection fraction by MUGA (required only if deemed clinically necessary for assessment) Other: No medical condition that would preclude protocol therapy: No severe diabetes No active ulcer disease No significant psychiatric disease No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Curatively treated Stage I cervical carcinoma Pretreatment mammogram and chest x-ray completed no more than 3 months preoperatively; blood/body fluid analyses to determine eligibility completed within 14 days prior to registration; prestudy bone scan completed within 12 weeks prior to registration and/or within 4 weeks prior to surgery

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No prior hormonal therapy (except for up to 14 days of tamoxifen stopped prior to registration) Prior estrogen- and/or progesterone-containing hormone preparations for nononcologic therapy allowed, but must be discontinued prior to registration Postmenopausal estrogen therapy should be discontinued in all patients at the time of diagnosis of breast cancer Radiotherapy: Postoperative chest wall and/or regional lymph node irradiation allowed for mastectomy patients (at discretion of the physician) either prior to registration or on protocol for any of the following: Tumor greater than 5 cm in diameter 4 or more positive nodes Extranodal extension of tumor into the axillary fat No radiotherapy for any other reason in mastectomy patients Postoperative radiotherapy either prior to registration, during tamoxifen, or after completion of chemotherapy required for lumpectomy patients Radiotherapy must be completed (if it is to be given before chemotherapy) prior to registration No immediate radiotherapy after randomization to chemotherapy Surgery: Radical, modified radical, or breast-sparing surgical procedure with at least a level I and II axillary dissection and analysis of at least 6 nodes required within 12 weeks prior to registration Lumpectomy must include: Total excisional biopsy with rim of normal breast tissue Microscopically negative margins Level I and II axillary dissection Tumor no more than 5 cm in greatest diameter Clinical and mammographic examination demonstrating absence of multicentric lesions Type of surgery, number of nodes examined, number of positive nodes, and size of the primary tumor (size of the largest tumor if more than 1 mass) must be recorded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1558 (Actual)
Dates: Start 1989-05; Primary Completion 2005-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | eight years
Overall survival | eight years
Toxicity/morbidity of treatment | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kathy S. Albain, MD, Study Chair — Loyola University; Charles D. Cobau, MD, Study Chair — Flower Hospital Cancer Center; James N. Ingle, MD, Study Chair — Mayo Clinic; Ellis G. Levine, MD, Study Chair — Roswell Park Cancer Institute; Kathleen I. Pritchard, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre

REFERENCES:
- [Background] Hershman DL, Unger JM, Barlow WE, Hutchins LF, Martino S, Osborne CK, Livingston RB, Albain KS. Treatment quality and outcomes of African American versus white breast cancer patients: retrospective analysis of Southwest Oncology studies S8814/S8897. J Clin Oncol. 2009 May 1;27(13):2157-62. doi: 10.1200/JCO.2008.19.1163. Epub 2009 Mar 23. PMID 19307504
- [Background] Hershman D, Unger J, Barlow W, et al.: Treatment quality and outcome of African American vs. European American breast cancer patients: retrospective analysis of Southwest Oncology Group studies S8814/S8897. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-3049, S140-1, 2006.
- [Background] Albain KS, Green SR, Lichter AS, Hutchins LF, Wood WC, Henderson IC, Ingle JN, O'Sullivan J, Osborne CK, Martino S. Influence of patient characteristics, socioeconomic factors, geography, and systemic risk on the use of breast-sparing treatment in women enrolled in adjuvant breast cancer studies: an analysis of two intergroup trials. J Clin Oncol. 1996 Nov;14(11):3009-17. doi: 10.1200/JCO.1996.14.11.3009. PMID 8918499
- [Result] Albain K, Barlow W, Shak S, et al.: Prognostic and predictive value of the 21-gene recurrence score assay in postmenopausal, node-positive, ER-positive breast cancer (S8814, INT0100). [Abstract] Breast Cancer Res Treat 106 (1): A-10, 2007.
- [Result] Albain K, Barlow W, O'Malley F, et al.: Concurrent (CAFT) versus sequential (CAF-T) chemohormonal therapy (cyclophosphamide, doxorubicin, 5-fluorouracil, tamoxifen) versus T alone for postmenopausal , node-positive, estrogen (ER) and/or progesterone (PgR) receptor-positive breast cancer: mature outcomes and new biologic correlates on phase III intergroup trial 0100 (SWOG-8814). [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-37, 2004.
- [Result] Albain KS, Green SJ, Ravdin PM, et al.: Adjuvant chemohormonal therapy for primary breast cancer should be sequential instead of concurrent: initial results from intergroup trial 0100 (SWOG-8814). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-143, 2002.
- [Result] Albain K, Green S, Ravdin P, et al.: Overall survival after cyclophosphamide, adriamycin, 5-Fu, and tamoxifen (CAFT) is superior to T alone in postmenopausal, receptor(+), node(+) breast cancer: new findings from phase III Southwest Oncology Group intergroup trial S8814 (INT-0100). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-94, 24a, 2001.
- [Result] Ravdin P, Green S, Albain K, et al.: Initial report of the SWOG biological correlative study of c-erB-2 expression as a predictor of outcome in a trial comparing adjuvant CAF T with tamoxifen (T) alone. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A374, 97a, 1998.
- [Result] Albain K, Green S, Osborne K, et al.: Tamoxifen (T) versus cyclophosphamide, adriamycin and 5-FU plus either concurrent or sequential T in postmenopausal, receptor(+), node(+) breast cancer: a Southwest Oncology Group phase III intergroup trial (SWOG-8814, INT-0100). [Abstract] Proceedings of the American Society of Clinical Oncology 16: A-450, 128a, 1997.
- [Derived] Pusztai L, Hoag JR, Albain KS, Barlow WE, Stemmer SM, Meisner A, Hortobagyi GN, Shak S, Rae JM, Baehner R, Sharma P, Kalinsky KM. Development and Validation of the RSClinN+ Tool to Predict Prognosis and Chemotherapy Benefit for Hormone Receptor-Positive, Node-Positive Breast Cancer. J Clin Oncol. 2025 Mar 10;43(8):919-928. doi: 10.1200/JCO-24-01507. Epub 2024 Dec 2. PMID 39621968
- [Derived] Speers CW, Symmans WF, Barlow WE, Trevarton A, The S, Du L, Rae JM, Shak S, Baehner R, Sharma P, Pusztai L, Hortobagyi GN, Hayes DF, Albain KS, Godwin A, Thompson A. Evaluation of the Sensitivity to Endocrine Therapy Index and 21-Gene Breast Recurrence Score in the SWOG S8814 Trial. J Clin Oncol. 2023 Apr 1;41(10):1841-1848. doi: 10.1200/JCO.22.01499. Epub 2023 Jan 17. PMID 36649570
- [Derived] Albain KS, Barlow WE, Ravdin PM, Farrar WB, Burton GV, Ketchel SJ, Cobau CD, Levine EG, Ingle JN, Pritchard KI, Lichter AS, Schneider DJ, Abeloff MD, Henderson IC, Muss HB, Green SJ, Lew D, Livingston RB, Martino S, Osborne CK; Breast Cancer Intergroup of North America. Adjuvant chemotherapy and timing of tamoxifen in postmenopausal patients with endocrine-responsive, node-positive breast cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Dec 19;374(9707):2055-2063. doi: 10.1016/S0140-6736(09)61523-3. Epub 2009 Dec 10. PMID 20004966